CLINICAL TRIAL: NCT01342237
Title: Tandem High Dose Chemotherapy and Autologous Stem Cell Rescue for High Risk Pediatric Brain Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Hyo Seop Ahn, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-SCT-1102
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Brain Tumors
Keywords: Brain tumors; Stem cell transplantation; topotecan; thiotepa; carboplatin; melphalan; etoposide
MeSH Terms: conditions — Brain Neoplasms | interventions — Topotecan; Thiotepa; Carboplatin; Melphalan; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- topotecan (Experimental)
  Interventions: Drug: HDCT 1(TTC), HDCT2(MEC)

INTERVENTIONS:
Drug: HDCT 1(TTC), HDCT2(MEC) — 1. TTC Topotecan (2 mg/m2 once daily i.v. on days -8, -7, -6, -5, -4) Thiotepa (300 mg/m2 once daily i.v on days -8, -7, -6) Carboplatin (500 mg/m2 once daily i.v on days -5, -4, -3) (max. 700 mg/day)
  2. MEC Melphalan (140 mg/m2 once daily i.v on day -7, 70 mg/m2 once daily i.v on day -6) Etoposide (200 mg/m2 once daily i.v on days -8, -6) Carboplatin (350 mg/m2 once daily i.v on days -8, -7, -6, -5)
  Other Names: Topotecan; Thiotepa; Carboplatin; Melphalan; Etoposide

SUMMARY:
The investigators plan to improve event free survival rate and reduce treatment related toxicities of pediatric patients with high risk/recurrent CNS tumors by administrating tandem high dose chemotherapy and autologous stem cell rescue.

DETAILED DESCRIPTION:
High risk/recurrent central nervous system (CNS) tumors have a poor prognosis so that tandem high dose chemotherapy (HDCT) with hematopoietic progenitor stem cell rescues has been chosen as potentially curative therapy. Many institutions have used carboplatin, thiotepa, etoposide (CTE) for conditioning regimen of 1st HDCT and cyclophosphamide, melphalan (CM) for conditioning regimen of 2nd HDCT. Our institution applied this regimen to the 38 pediatric patients with high risk brain tumor since 1996. Although the 3 year overall survival rate and event free survival rate were improved to 69% and 47.9%, respectively, the results showed relatively high treatment related mortality (TRM) rate of 21%. Toxicity of this tandem regimen was also reported as being high up to 32% in other researches as well so that this regimen is considered not feasible due to toxicity. In this study, the investigators plan to improve event free survival rate and reduce treatment related toxicities of pediatric patients with high risk/recurrent CNS tumors by administrating tandem high dose chemotherapy and autologous stem cell rescue with topotecan, thiotepa, carboplatin (TTC) for 1st HDCT and melphalan, etoposide, carboplatin (MEC) for 2nd HDCT.

ELIGIBILITY:
Inclusion Criteria:

1. High risk pediatric brain tumors Newly diagnosed medulloblastoma, CNS PNET, ATRT, Choroid plexus carcinoma, pineoblastoma with residual tumor over 1.5cm2 after operation or with leptomeningeal seeding at diagnosis
2. All high grade or malignant brain tumor, age < 3 years
3. Recurrent embryonal brain tumors, recurrent CNS germ cell tumor
4. Age : no limitation
5. Performance status : ECOG 0-2.
6. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.

   Heart: a shortening fraction ≥ 28%. Liver: total bilirubin < 2 ⅹ upper limit of normal; ALT < 3 ⅹ upper limit of normal. Kidney: creatinine < 2 ⅹ normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
7. Patients must lack any active viral infections or active fungal infection.
8. Patients (or one of parents if patients age < 20) should sign informed.

Exclusion Criteria:

1. Patients who do not reach partial response prior to high dose chemotherapy.
2. Pregnant or nursing women.
3. Malignant (except brain tumor) or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
4. Psychiatric disorder that would preclude compliance.
5. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate event free survival rate | 1 month
  To evaluate event free survival rate after high dose chemotherapy and autologous stem cell rescue in pediatric patients with high risk brain tumor

SECONDARY OUTCOMES:
To evaluate treatment related mortality | 1, 3, 6, 12 month
To evaluate the incidence and severity of toxicity | 1, 3, 6, 12 month
To evaluate overall survival rate and relapse rate | 1, 3, 6, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea